CLINICAL TRIAL: NCT00281320
Title: A Randomized, Parallel Group, Multiple Dose, 6-Week Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Asenapine in Elderly Subjects With Psychosis.
Brief Title: Study of Asenapine in Elderly Subjects With Psychosis (A7501021)(P05717)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05717; A7501021
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine 2-10 mg BID (Experimental): Dose titration from 2 mg to 5 mg to 10 mg twice daily (BID)
  Interventions: Drug: Asenapine
- Asenapine 5-10mg BID (Experimental): Dose titration from 5 mg to 10 mg BID
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Asenapine — Asenapine 2 mg twice daily (BID) on Days 1 and 2, 5 mg BID on Days 3 and 4, followed by 10 mg BID on Day 5 through the end of the trial (Week 6); or Asenapine 5 mg BID on Days 1 to 4 followed by 10 mg BID on Day 5 through the end of the trial (Week 6).
  Other Names: Saphris

SUMMARY:
This study evaluates the safety and tolerability of Asenapine in elderly patients with psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Elderly subjects with psychosis

Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant

medical condition.

* Have an established diagnosis of dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Result] Dubovsky SL, Frobose C, Phiri P, de Greef R, Panagides J. Short-term safety and pharmacokinetic profile of asenapine in older patients with psychosis. Int J Geriatr Psychiatry. 2012 May;27(5):472-82. doi: 10.1002/gps.2737. Epub 2011 Jul 13. PMID 21755540

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine 2-10 mg Twice Daily (BID): Asenapine 2 mg twice daily (BID) on Days 1 and 2, 5 mg BID on Days 3 and 4, followed by 10 mg BID on Day 5 through the end of the trial (Week 6)
- Asenapine 5-10 mg BID: Asenapine 5 mg BID on Days 1 to 4 followed by 10 mg BID on Day 5 through the end of the trial (Week 6)
Period: Overall Study
Arm/Group | Asenapine 2-10 mg Twice Daily (BID) | Asenapine 5-10 mg BID
Started | 61 | 61
Completed | 36 | 40
Not Completed | 25 | 21
Not completed — Adverse Event | 12 | 9
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Asenapine 2-10 mg BID: Asenapine 2 mg twice daily (BID) on Days 1 and 2, 5 mg BID on Days 3 and 4, followed by 10 mg BID on Day 5 through the end of the trial (Week 6)
- Asenapine 5-10 mg BID: Asenapine 5 mg twice daily (BID) on Days 1 to 4 followed by 10 mg BID on Day 5 through the end of the trial (Week 6)
- Total: Total of all reporting groups
Arm/Group | Asenapine 2-10 mg BID | Asenapine 5-10 mg BID | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (4.6) | 72.0 (5.8) | 71.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 47 | 88
  Male | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: Participants who experienced treatment-emergent adverse events, defined as newly reported events after baseline or events reported to have worsened in severity since baseline (from the date of informed consent to the last dose day + 7 days for non-serious adverse events and 30 days for serious adverse events).
Time Frame: Up to Day 42 (treatment period)
Population: Per protocol
Measure: Number; unit: Participants
Groups:
- Asenapine 2-10 mg Twice Daily (BID): Asenapine 2 mg twice daily (BID) on Days 1 and 2, 5 mg BID on Days 3 and 4, followed by 10 mg BID on Days 5 through the end of the trial (Week 6)
- Asenapine 5-10 mg BID: Asenapine 5 mg BID on Days 1 to 4 followed by 10 mg BID on Days 5 through the end of the trial (Week 6)
Arm/Group | Asenapine 2-10 mg Twice Daily (BID) | Asenapine 5-10 mg BID
Number analyzed (Participants) | 61 | 61
Participants | 44 | 44

2. Primary Outcome: Number of Participants Who Discontinued Because of an Adverse Event
Description: Discontinuations due to treatment-emergent adverse events starting on or after Day1 and up to 7 days after study medication stop date (30 days for serious adverse events).
Time Frame: up to 30 days after study medication stop date
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Asenapine 2-10 mg Twice Daily (BID) | Asenapine 5-10 mg BID
Number analyzed (Participants) | 61 | 61
participants | 12 | 9

3. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis, Tmax
Description: Tmax defined as time to peak concentration.
Time Frame: Day 4 or 8
Population: All-Subjects-Pharmacokinetically-Evaluable Group defined as all subjects for which at least one pharmacokinetic parameter could be calculated and who did not have any protocol violations interfering with pharmacokinetics.
Measure: Median (Full Range); unit: hours
Groups:
- Asenapine 5mg BID Day 4: Pharmacokinetic parameter of asepanine for Day 4.
- Asenapine 10mg BID Day 8: Pharmacokinetic parameter of asepanine for Day 8.
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 87 | 60
hours | 1.00 [0.417 to 4.23] | 1.06 [0.417 to 4.08]

4. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis,Cmax
Description: Cmax defined as peak concentration.
Time Frame: Day 4 or 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 87 | 60
ng/mL | 6.01 (3.89) | 10.3 (6.71)

5. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis , Dn-Cmax
Description: dn-Cmax is defined as dose normalized peak concentration.
Time Frame: Day 4 or 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 87 | 60
ng/mL/mg | 1.20 (0.778) | 1.03 (0.671)

6. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis, Cmin
Description: Cmin defined as pre-dose concentration.
Time Frame: Day 4 or 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Asenapine 5mg BID Day 4: Pharmacokinetic parameters of asepanine for Day 4.
- Asenapine 10mg BID Day 8: Pharmacokinetic parameters of asepanine for Day 8.
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 86 | 60
ng/mL | 2.28 (1.87) | 4.06 (2.70)

7. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis, AUC 0-12
Description: AUC 0-12 defined as area-under-the-curve from zero to time point 12 hours.
Time Frame: Day 4 or 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Asenapine 5mg BID Day 4: Pharmacokinetic parameter of asenapine for Day 4.
- Asenapine 10mg BID Day 8: Pharmacokinetic parameter of asenapine for Day 8.
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 87 | 60
ng*h/mL | 38.6 (21.1) | 70.3 (41.8)

8. Primary Outcome: Pharmacokinetics of Asenapine up to Doses of 10 mg BID in Elderly Subjects With Psychosis, Dn-AUC 0-12
Description: dn-AUC 0-12 defined as dose-normalized area-under-the-curve from zero to time point 12 hours.
Time Frame: Day 4 or 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL/mg
Arm/Group | Asenapine 5mg BID Day 4 | Asenapine 10mg BID Day 8
Number analyzed (Participants) | 87 | 60
ng*h/mL/mg | 7.72 (4.22) | 7.03 (4.18)

ADVERSE EVENTS:
Arm/Group | Asenapine 2-10mg BID | Asenapine 5-10mg BID
Serious Adverse Events (participants affected / at risk) | 6/61 | 3/61
Other Adverse Events (participants affected / at risk) | 21/61 | 21/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 2-10mg BID (N=61) | Asenapine 5-10mg BID (N=61)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 2-10mg BID (N=61) | Asenapine 5-10mg BID (N=61)
Asthenia (General disorders) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 5 (7)
Dizziness (Nervous system disorders) | 4 (4) | 2 (3)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Parkinsonism (Nervous system disorders) | 1 (1) | 5 (6)
Somnolence (Nervous system disorders) | 5 (6) | 3 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 7 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will provide manuscripts, abstracts, or the full text of any other intended disclosure to the sponsor at least 30 days prior to submission for publication or other disclosure. If any patent action is required to protect intellectual property rights, Institution agrees to delay the disclosure for a period not to exceed and additional 60 days. Institution will, on request, remove any previously undisclosed Confidential Information (other than study results) before disclosure.